CLINICAL TRIAL: NCT06175897
Title: Effects of STN Deep Brain Stimulation on Cognition and Brain Networks in Parkinson's Disease Patients Analyzed Based on EEG and Functional Near-infrared Spectroscopy
Brief Title: Effects of STN DBS on Cognition and Brain Networks in PD Patients Analyzed Based on EEG and fNIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhiqi Mao (Other)
Responsible Party: Sponsor-Investigator, Zhiqi Mao, Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChinaPLAGH-ZH
Record Dates: First submitted 2023-11-28; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Parkinson's Disease; Executive Function; Electroencephalogram; Functional Near - Infrared Spectroscopy
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical group (Experimental): Undergoing DBS
  Interventions: Procedure: Deep Brain Stimulation
- control group (Sham Comparator): Undergoing non-DBS
  Interventions: Procedure: non-Deep Brain Stimulation

INTERVENTIONS:
Procedure: Deep Brain Stimulation — An elaborate target/trajectory planning and a precise image fusion of MRI and stereotactic CT scanning are performed before surgery. After microelectrode recording, two sets of quadripolar DBS leads (contact interval is 0.5mm) will be inserted into the dorsolateral part of bilateral STN nuclei separately. Subsequently, an implantable pulse generator will be connected via extension wires and implanted at the left/right subclavicular area subcutaneously.
  Device: STN-DBS devices DBS electrode: 3389 (Medtronic, Minneapolis, MN, USA) or L301 (PINS Medical, Beijing, China) or 1200 (SceneRay, Suzhou, China); Extension wire: 37086 (Medtronic, Minneapolis, MN, USA) or E202 (PINS Medical, Beijing, China) or 1340/SR1341 (SceneRay, Suzhou, China); Implantable pulse generator: ACTIVA PC/RC (Medtronic, Minneapolis, MN, USA) or G102/G102R (PINS Medical, Beijing, China) or 1180/SR1101 (SceneRay, Suzhou, China).
  Arms: surgical group
Procedure: non-Deep Brain Stimulation — Patients with PD were given their original drug dose and did not receive DBS.
  Arms: control group

SUMMARY:
In recent years, deep brain stimulation (DBS) has become the primary treatment for patients with medically uncontrolled Parkinson's disease (PD). Nevertheless, previous studies have shown that it has been controversial whether DBS-subthal amic nucleus (STN) has facilitated or impaired cognitive function in patients with PD. The etiology of the effect of DBS on the single cognitive domain, executive function, has yet to be clarified. Previous clinical studies in which DBS was performed in patients with PD have been performed under the Stroop effect. TMT (Trail Making Test A and B) cognitive tests and simultaneous acquisition of brain function data by electroencephalograph-functional near-infrared spectroscopy (EEG-fNIRS) have yet to be reported.

To investigate the effect of DBS-STN on executive function in PD patients and whether there are differences at baseline, 1-month postoperative (DBS-on), 6 months postoperative follow-up, and 12 months postoperative follow-up. Under the condition of electroencephalograph-functional near-infrared spectroscopy (EEG-fNIRS) bimodal technology fusion, The investigators allow PD patients to operate the test of executive function (Stroop/TMT), real-time monitoring of cranial neurophysiology-oxygenation signals, and explore the changes of the brain function network of PD patients, and hope to achieve the following objectives through objective and scientific-technological means: (1) quantify the cognitive function of PD patients through EEG-fNIRS technology and possible trends of changes; (2) explain whether executive functions differ at the level of brain functional network connectivity between surgical and conservative treatments and whether the differences have interaction effects with treatment duration and treatment modalities, as well as analyze their simple effects; (3) To minimize artificial confounders of short-term learning effects and testers common to previous neurocognitive psychobehavioral tests; (4) To explore the mechanism of DBS on the changes of cortical brain networks in PD patients, to avoid or reduce the interference of surgery on cognitive functions, and to provide a theoretical basis for treating personalized surgical plans.

DETAILED DESCRIPTION:
In recent years, deep brain electrical stimulation (DBS) has become a primary treatment for improving clinical symptoms in Parkinson's disease (PD) patients with predominantly motor slowing after poor drug effects from conventional drug therapy medications or after the progression of the disease. However, previous studies have been controversial in examining whether DBS-STN promotes or impairs cognitive function in patients with PD. Previous studies have found that DBS may affect executive function in patients with PD and that specific brain regions are closely related to executive function. In this study, the investigators used electroencephalograph-functional near-infrared spectroscopy (EEG-fNIRS) to obtain brain network connectivity in subjects and to explore the possible relationship between executive function and brain network connectivity in patients with Parkinson's disease. To explore the possible brain network connectivity affecting execution in DBS-STN and to predict postoperative executive function in PD patients in DBS.

Among the single cognitive domains impaired, executive function impairment is the most common, accounting for more than 70% of the cases, and impairment of attention, working memory, and visuospatial ability are also more common. Impaired executive function is the most characteristic cognitive impairment in PD patients, which is related to the disruption of the integrity of the frontal-striatal loops, designing a wide range of functional brain regions, such as the frontal lobe, parietal lobe, cingulate gyrus, thalamus, substantia nigra, and so on, and clinically manifested as impaired cognitive flexibility, planning, concept formation, working memory, and learning ability. Executive dysfunction can seriously affect patients' social behavior, especially when performing more complex tasks that require the integration of multiple steps in a particular order.

Previous studies have found that brain network connectivity in specific brain regions is closely related to cognitive function, for example, there have been many clinical studies based on functional MRI blood oxygenation signals, but because of the poor immunity to electromagnetic interference, patients with implanted electrodes have to be DBS-off in order to do the MRI. Because of poor anti-motor interference, only some motor imagery and simple finger movements can be acquired under the DBS-off condition for functional MRI, and functional MRI has been an important issue limiting cognitive neuroscience research due to its low temporal resolution and its inability to monitor in real-time the changes of cortical brain blood oxygenation signals in the task paradigm.

Therefore, this study plans to design a multicenter, prospective, randomized, parallel-controlled equipotent clinical trial, which innovatively combines electroencephalography (EEG) with high temporal resolution and functional near-infrared spectroscopy (fNIRS) with a high spatial resolution to monitor cortical oxygenation signals in real-time, so that the brain electrophysiological and blood oxygenation signals can be acquired in real-time during a test of executive function (Stroop/TMT). The real-time measurement and evaluation of cognitive function by synchronously acquiring electrophysiological and oxygenation signaling changes in the brain while the patient is performing the executive function test (Stroop/TMT) and obtaining real-time EEG-fNIRS brain network data during the executive function test has always been a higher-order field of cognitive function research. The present study investigated the mechanisms of executive function impairment in PD patients and whether DBS-STN affects the brain network mechanisms of executive function. It is hoped to (1) quantify cognitive function and possible trends in cognitive functioning in PD patients by EEG-fNIRS technique, (2) Explain whether there are differences in executive function at the level of brain functional network connectivity between surgical and conservative treatments and whether there are interaction effects of the differences with the duration of treatment and the treatment modality as well as to analyze their simple effects, (3) To minimize artificial confounders of short-term learning effects and testers familiar with previous neurocognitive psychobehavioral tests, (4) To explore the mechanism of DBS on the changes of cortical brain networks in PD patients, to avoid or reduce the interference of surgery on cognitive functions, and to provide a theoretical basis for treating personalized surgical plans.

In this study, the investigators planned to design a multicenter, prospective, randomized, parallel-controlled clinical trial. A total of 80 patients were randomly assigned to the DBS-STN group. The DBS treatment group, with the non-DBS treatment group, routinely DBS-on at 1 month postoperatively. The conservative treatment routinely on oral medication and the data on patients' brain function was collected by the simultaneous EEG-fNIRS bimodal technique in combination with cognitive testing (Stroop/TMT) at baseline, 1 month after DBS (DBS-on), and at 6 months/12 months after DBS, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary PD whose diagnosis meets "China's Diagnostic Criteria for Parkinson's Disease" issued in 2016.
2. Disease duration: In principle, PD patients with disease duration ≥5 years, patients with disease duration <5 years but meeting the clinical confirmation criteria for primary PD, with confirmation of surgical indications, the duration of the disease can be relaxed to 4 years, PD patients with predominantly tremor, with unsatisfactory improvement of tremor by standardized drug therapy and severe tremor affecting the patient's quality of life, the duration of the disease can be relaxed to 3 years after evaluation.
3. Patients who have received levodopa medication with good efficacy and ≥30% improvement of symptoms in dopamine shock test.
4. Significant decrease in the efficacy of drug therapy, intolerable motor complications, and drug side effects.
5. Disease severity: In patients with symptomatic fluctuation of the "on-off" phenomenon, the Hoehn-Yahr stage of the off phase is 2.5-4.0.
6. Age: The age of patients undergoing surgery is usually <75 years old, and if the patient's physical condition is good, the age limit can be appropriately relaxed.
7. Those who agree to undergo evaluation and can cooperate to complete the follow-up.

Exclusion Criteria：

1. Have significant cognitive dysfunction.
2. Have a psychiatric disorder such as severe depression, anxiety, or schizophrenia.
3. Have underlying severe diseases that cannot tolerate surgery or affect post-operative survival.
4. The disease has progressed to the terminal stage, and the patient is entirely unable to take care of himself/herself and is bedridden.
5. Those with abnormal intracranial lesions and contraindications to MRI scanning, such as those with metal implants, claustrophobia, etc.
6. Parkinson's disease syndrome and Parkinson's superimposed syndrome caused by other reasons.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in EEG-fNIRS performance | up to 1 month (DBS-on) ,6 months，12 months
  To explore the differences in cognitive brain network changes in PD patients by using EEG-fNIRS photofusion technology. The EEG-fNIRS bimodal brain network of PD patients were constructed, and the network characteristic indexes, such as node degree, characteristic path length, and clustering coefficient, were counted. The cognitive differences of PD patients were interpreted by the actual physiological state represented by the brain network feature indicators, for example, a high node entry degree means high information inflow in the brain area where the node is located, short feature path length means high efficiency of whole-brain information transfer in the patient, and large clustering coefficient means high degree of modularity in the brain area of the PD patient. These characteristic indexes can better reflect PD patients' cognitive state and change differences.

SECONDARY OUTCOMES:
Change in Stroop scores | up to 1 month (DBS-on), 6 months, 12 months
  Stroop A, B, and C elapsed time per card, number of correct (timing accurate to 0.01 s).
  The metrics reflecting the amount of interference (Stroop interference effect, SIE) include:
  SIE elapsed time = card C elapsed time - card B elapsed time; SIE correct number = card B correct number - card C correct number. The larger the SIE is, the lower the interference suppression effect is, and the more serious the impairment of executive function is.
  The indexes observed in this study include the number of correct and elapsed times of cards A, B, and C, the number of elapsed time and correct number of SIE, the elapsed time of cards (C-A-B), the rate of increase of elapsed time (C-B)/A, the rate of decrease of correct number (B-C)/A, and the elapsed time/correct number of each card.
Change in Trail Making Test A and B scores | up to 1 month (DBS-on), 6 months, 12 months
  TMT-A, and TMT-B recording indicators include: TMT-A elapsed time number (timing accurate to 0.01s); TMT-B elapsed time number (timing accurate to 0.01s); Number of TMT-A and TMT-B error connection reminders, number of pen lifts; Interference Error Coefficient (IE): (TMT-A - TMT-B) / TMT-A
Change in Mini-mental State Examination scores | up to 1 month (DBS-on), 6 months, 12 months
  Mini-mental State Examination (MMSE) will be used to evaluate the general cognitive function. MMSE ranges from 0 to 30, and a higher value represents a better outcome.
Change in Neuropsychiatric Inventory (NPI) scores | up to 1 month (DBS-on), 6 months, 12 months
  The Neuropsychiatric Inventory will be used to measure neuropsychiatric symptoms. It ranges from 0 to 144, and higher value represents a worse outcome.
Change in Activities of Daily Living scores | up to 1 month (DBS-on), 6 months, 12 months
  Activities of Daily Living (ADL) scale will be used to assess the change of life quality. It ranges from 20 to 80. The "20" represents normal life ability and the higher score presents the worse life ability.
Change in Montreal Cognitive Assessment scores | up to 1 month (DBS-on), 6 months, 12 months
  Montreal Cognitive Assessment (MoCA) will be used to evaluate the general cognitive function. MoCA ranges from 0 to 30, and higher value represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqi Mao, PhD, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China